CLINICAL TRIAL: NCT02050620
Title: A Pilot Study to Examine the Association Between Self-Reported Exercise Behavior and Short-Term Patient Outcomes in Women Undergoing Radiation Treatment for Operable Breast Cancer
Brief Title: Self-Reported Exercise Behavior and Short-Term Patient Outcomes in Women Undergoing Radiation Treatment for Operable Breast Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050716
Record Dates: First submitted 2014-01-23; First posted 2014-01-31 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer, exercise and quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Using an observational prospective design, potential subjects will be identified and screened for eligibility via medical record review of breast cancer patients scheduled for radiation therapy at Duke Radiation Oncology Clinic. Subjects who agree to participate will be asked to complete study questionaires prior to the start of radiation therapy and again during the last week of therapy.

DETAILED DESCRIPTION:
Exercise behavior will be defined as patient reported mean total minutes (frequency x duration) of mild, moderate, and vigorous-intensity physical exercise per week over the past month at baseline (prior to enrollment in the study). In addition we will collect patient reported mean total minutes per week of mild, moderate, and vigorous-intensity physical exercise over the course of radiation therapy.Baseline characteristics including demographic data (age, education, employment) as well as BMI, waist to hip ratio, and health comorbidities (including smoking status, cardiovascular disease, and diabetes) will also be collected. BMI and health comorbidities will be extracted from the chart. Patient-Reported Outcomes will include QOL, fatigue, depression, pain and sleep. QOL will be assessed using the Functional Assessment of Cancer Therapy (FACT) scale developed for the assessment of patient symptoms and QOL in cancer patients. Fatigue will be assessed using the 13-item FACT-fatigue scale for the assessment of fatigue in cancer patients.Skin toxicity will be defined as radiation dermatitis, pruritus, and pain.

Lymphedema will be assessed by measuring limb girth. Measurements will be taken by first marking both limbs while patient is lying supine, starting at the ulnar styloid at 5cm intervals on the length of the arms. The diameter of the limb will then be measured at these markings. Based on these measurements, the affected limb will be compared to the unaffected limb. Range of motion will be defined as reduced abduction compared to the contralateral shoulder . All measurements will be taken with a goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Women with a biopsy-proven diagnosis of ductal carcinoma in situ or invasive breast carcinoma
* Definitive radiation treatment planned to the chest and/or regional nodes
* 18 years of age or older
* Signed study-specific informed consent

Exclusion Criteria:

* Significant mental disorders making informed consent difficult or mental impairment leading to inability to cooperate
* Karnofsky Performance Status (KPS) < 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with biopsy proven ductal carcinoma in situ or invasive breast carcinoma scheduled to receive definitive treatment in the Department of Radiation Oncology at Duke will be potentially eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To measure in composite the association between self reported exercise behaviour and patient reported outcomes of quality of life. | 24 months
  Quality of life outcomes will be measured by patient self reported levels of fatigue, sleep, pain and depression. Patient-Reported Outcomes will include QOL, fatigue, depression, pain and sleep. QOL will be assessed using the Functional Assessment of Cancer Therapy (FACT) scale. Fatigue will be assessed using the 13-item FACT-fatigue scale. Beck depression inventory (BDI) will be used to evaluate for underlying depressive symptoms. We will use the revised version (BDI-II) and the scores will range from 0 (no depression) to 63 (severe depression) (Beck et al., 1996) Pain will be assessed using the previously validated shortened Brief Pain Inventory (BPI) (Cleeland & Ryan, 1994). Sleep will be measured using the previously validated Pittsburgh Sleep Inventory (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989).

SECONDARY OUTCOMES:
To measure in composite the association between self-reported exercise behavior and acute radiation related toxicities. | 24 months
  Acute radiation related toxicities will include assessments of radiation dermatitis , range of motion and lymphedema.Skin toxicity will be defined as radiation dermatitis, pruritus, and pain. It will be evaluated using the National Cancer Institute Common Terminology Criteria of Adverse Events v4.0 (NCI, 2010).
  Lymphedema will be assessed by measuring limb girth. Measurements will be taken by first marking both limbs while patient is lying supine, starting at the ulnar styloid at 5cm intervals on the length of the arms. The diameter of the limb will then be measured at these markings. Based on these measurements, the affected limb will be compared to the unaffected limb. Lymphedema will be classified according to the American System: Mild 1.5-3.0 cm; Moderate 3.1-5.0 cm; Severe > 5.0 cm.(Markowski, Wilcox, & Helm, 1981) Range of motion will be defined as reduced abduction compared to the contralateral shoulder . All measurements will be taken with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Janet K Horton, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States